CLINICAL TRIAL: NCT03851770
Title: NEURO-LARYNX:Laryngeal Motor Evoked-potentials as a Biomarker of Vagus Nerve Stimulation
Brief Title: Laryngeal Motor Evoked-potentials as a Biomarker of Vagus Nerve Stimulation in Epileptic Patients
Acronym: NEURO-LARYNX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/07NOV/416
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Patients participating will be asked to come to the Neurophysiology Department of Saint Luc Clinic to peform the laryngeal evoked motor potential.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- refractory epilepsy patients (Other): All patients belong to the refractory epilepsy group. Intervention: Characterization of Vagus nerve stimulation: Evoked potentials (EP) are recorded using an EEG/EP digital acquisition system
  Interventions: Other: Characterization of Vagus nerve stimulation

INTERVENTIONS:
Other: Characterization of Vagus nerve stimulation — Characterization of Vagus nerve stimulation induced larynx evoked motor potential. Patients participating in the study will be asked to come to perform the experiment (duration maximum 1 hour) at the Neurophysiology Department of Saint Luc .

SUMMARY:
The goal of this study is to record and characterize larynx evoked motor potentials induced by vagus nerve stimulation. This study will include 10 adult patients implanted with a Vagus nerve stimulator, followed at the Center for Refractory Epilepsy at Cliniques St Luc. The inclusion criteria are: (1) patient aged between 18 and 65 years ; (2) cervical VNS device (Cyberonics, Houston, TX, USA) implanted for at least 6 months, (3) normal electrode impedance of the electrode. Exclusion criteria are (1) presence of a concomitant laryngeal pathology or recurrent laryngeal nerve damage, independent from VNS ; (2) important VNS side effects reported by the patient, such as severe dyspnea (grade III-IV) or severe pain in the neck/ear region.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18 and 65 years
* Vagus nerve stimulation implanted for at least 6 months
* No impedance issues with the VNS electrode

Exclusion Criteria:

* presence of a concomitant laryngeal pathology or RLN damage, independent from vagus nerve stimulation
* important side effects of the VNS reported by the patient such as dyspnea, pain in neck/ear region and gastrointestinal complaints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Laryngeal motor evoked potential (LMEP) | the LMEP is recorded for 60 minutes from the moment the patient arrives to the clinic to perform the test
  Characteristics of the laryngeal motor evoked potential Threshold : the mA of current output necessary for evoking the LMEP Latency : the time between the negative peak of the stimulation artifact and the first positive deflection of the LMEP Amplitude : the difference in μV between the lowest negative and the highest positive peak of the LMEP Duration : the time between the first positive deflection of LMEP and the return to the noise level Dose- response curve: the relation between increasing intensity of vagal nerve stimulation and amplitude of the LMEP

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires St Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided